CLINICAL TRIAL: NCT03894878
Title: Association Between Risk Scores for Genetic Variants and Percentage of Time in Therapeutic Range for Participants With Atrial Fibrillation, Deep Vein Thrombosis, and/or Intracardiac Thrombosis Taking Warfarin
Brief Title: Association Between Genetic Variant Scores and Warfarin Effect
Acronym: AWARE1
Status: Completed | Type: Observational
Sponsor: Cipherome, Inc. (Industry)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: C01-001 SC001
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Deep Vein Thrombosis; Intracardiac Thrombus; Pulmonary Embolism; Venous Thromboembolic Disease
Keywords: Warfarin; Coumadin; Pharmacogenomics; Pharmacogenetics; Adverse Drug Reactions; Bleeding/hemorrhaging
MeSH Terms: conditions — Atrial Fibrillation; Venous Thrombosis; Pulmonary Embolism; Drug-Related Side Effects and Adverse Reactions; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Sample collection:
  One 3 mL venous blood sample will be taken from each study participant and collected in EDTA tubes on the day of the one-time study visit, when the participant is reporting to the SCVH&HS laboratory to undergo INR testing per Anticoagulation Clinic protocol.
  This 3 mL venous blood sample will be taken from each study participant, in addition to the standard of care blood draw for INR. Each sample tube will be labeled with the protocol study number, along with the date and time of collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study objective is to determine whether there is an association between genetic variant risk scores and clinical outcomes (percent time in therapeutic range, time to reach therapeutic international normalized ratio (INR), INR ≥ 4, bleeding event, ischemic stroke, death) in participants taking warfarin for atrial fibrillation, deep vein thrombosis (DVT), pulmonary embolism (PE), and/or intracardiac thrombosis.

DETAILED DESCRIPTION:
It is anticipated that next generation genomic sequencing will identify rare genetic variants in ethnically diverse populations, which otherwise would not have been detected using commercially available warfarin tests. Furthermore, retrospective review of clinical outcomes (percent time in therapeutic range, time to reach therapeutic international normalized ratio (INR), INR ≥ 4, major bleeding event, ischemic stroke) of study participants will determine the clinical utility of genetic variant risk scores. Study outcomes will provide guidance on future directions for optimizing dosing algorithms for warfarin that combine pharmacogenetic principles with clinical dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Non-valvular atrial fibrillation
2. Deep venous thrombosis (DVT) and/or pulmonary embolism (PE) with no hypercoagulable condition
3. Non-valvular atrial fibrillation and DVT/PE (with no hypercoagulable condition)
4. Intracardiac thrombosis (i.e. apical thrombosis, atrial thrombosis, auricular thrombosis, mural thrombosis, and/or ventricular thrombosis)
5. Age 18-99 years
6. Signed informed consent

Exclusion Criteria:

1. Presence of a mechanical heart valve
2. Failure to provide signed informed consent
3. Known diseases that affects coagulation test results such as vitamin K deficiency, disseminated intravascular coagulopathy, Von Willebrand disease, hemophilia, liver failure, etc.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Participants with a known disease that predisposes them to bleeding will be excluded, since it will be a confounder (trying to link abnormal genetic variant risk score to bleeding).
  2. Participants taking medications or on a diet that increases bleeding propensity will also be excluded.
  3. Pediatric participants will be excluded from this study, since atrial fibrillation and/or venous thromboembolism are rare in this cohort.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Percent time in therapeutic range during initial 12 weeks of warfarin | 12 weeks
  Within the 12 weeks of treatment, this is the percentage of time that a given participant is within the therapeutic range (e.g. participant is in therapeutic range 75% of time/12 weeks of measurement)

SECONDARY OUTCOMES:
Time to reach therapeutic INR | 12 weeks
  Time needed to achieve first INR within the range of 2 to 3, provided that subsequent INR ≥ 7 days later was also within the range of 2 to 3
INR ≥ 4.0 during first 12 weeks of warfarin therapy | 12 weeks
  Time greater than the desired INR therapeutic range within the first 12 weeks of warfarin therapy
Ischemic stroke | 12 weeks
  Development of a clinical diagnosis of an ischemic stroke
Major bleeding event during first 12 weeks of warfarin therapy | 12 weeks
  Development of a major bleeding event during the first 12 weeks of warfarin therapy, diagnosed by a clinician
Clinically relevant non-major bleeding event during the first 12 weeks of warfarin therapy | 12 weeks
  Development of a clinically relevant non-major bleeding event during the first 12 weeks of warfarin therapy, diagnosed by a clinician

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Wang, MD, Principal Investigator — Santa Clara Valley Medical Center; Dayani Nualles-Percy, MD, Study Director — Santa Clara Valley Medical Center
Locations (1):
- Santa Clara Valley Medical Center, Santa Clara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colilla S, Crow A, Petkun W, Singer DE, Simon T, Liu X. Estimates of current and future incidence and prevalence of atrial fibrillation in the U.S. adult population. Am J Cardiol. 2013 Oct 15;112(8):1142-7. doi: 10.1016/j.amjcard.2013.05.063. Epub 2013 Jul 4. PMID 23831166
- [Background] Wysowski DK, Nourjah P, Swartz L. Bleeding complications with warfarin use: a prevalent adverse effect resulting in regulatory action. Arch Intern Med. 2007 Jul 9;167(13):1414-9. doi: 10.1001/archinte.167.13.1414. PMID 17620536
- [Background] Zareh M, Davis A, Henderson S. Reversal of warfarin-induced hemorrhage in the emergency department. West J Emerg Med. 2011 Nov;12(4):386-92. doi: 10.5811/westjem.2011.3.2051. PMID 22224125
- [Background] Johnson JA, Caudle KE, Gong L, Whirl-Carrillo M, Stein CM, Scott SA, Lee MT, Gage BF, Kimmel SE, Perera MA, Anderson JL, Pirmohamed M, Klein TE, Limdi NA, Cavallari LH, Wadelius M. Clinical Pharmacogenetics Implementation Consortium (CPIC) Guideline for Pharmacogenetics-Guided Warfarin Dosing: 2017 Update. Clin Pharmacol Ther. 2017 Sep;102(3):397-404. doi: 10.1002/cpt.668. Epub 2017 Apr 4. PMID 28198005
- [Background] Cavallari LH, Perera MA. The future of warfarin pharmacogenetics in under-represented minority groups. Future Cardiol. 2012 Jul;8(4):563-76. doi: 10.2217/fca.12.31. PMID 22871196
- [Background] https://www.bcbsks.com/CustomerService/Providers/MedicalPolicies/policies/policies/GeneticTesting_WarfarinDose_2017-09-01.pdf (Accessed July 22, 2019)
- [Background] Pirmohamed M, Burnside G, Eriksson N, Jorgensen AL, Toh CH, Nicholson T, Kesteven P, Christersson C, Wahlstrom B, Stafberg C, Zhang JE, Leathart JB, Kohnke H, Maitland-van der Zee AH, Williamson PR, Daly AK, Avery P, Kamali F, Wadelius M; EU-PACT Group. A randomized trial of genotype-guided dosing of warfarin. N Engl J Med. 2013 Dec 12;369(24):2294-303. doi: 10.1056/NEJMoa1311386. Epub 2013 Nov 19. PMID 24251363
- [Background] Kimmel SE, French B, Kasner SE, Johnson JA, Anderson JL, Gage BF, Rosenberg YD, Eby CS, Madigan RA, McBane RB, Abdel-Rahman SZ, Stevens SM, Yale S, Mohler ER 3rd, Fang MC, Shah V, Horenstein RB, Limdi NA, Muldowney JA 3rd, Gujral J, Delafontaine P, Desnick RJ, Ortel TL, Billett HH, Pendleton RC, Geller NL, Halperin JL, Goldhaber SZ, Caldwell MD, Califf RM, Ellenberg JH; COAG Investigators. A pharmacogenetic versus a clinical algorithm for warfarin dosing. N Engl J Med. 2013 Dec 12;369(24):2283-93. doi: 10.1056/NEJMoa1310669. Epub 2013 Nov 19. PMID 24251361
- [Background] Rosendaal FR, Cannegieter SC, van der Meer FJ, Briet E. A method to determine the optimal intensity of oral anticoagulant therapy. Thromb Haemost. 1993 Mar 1;69(3):236-9. PMID 8470047
- [Background] Schulman S, Kearon C; Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost. 2005 Apr;3(4):692-4. doi: 10.1111/j.1538-7836.2005.01204.x. PMID 15842354
- [Background] Lip GY. Intracardiac thrombus formation in cardiac impairment: the role of anticoagulant therapy. Postgrad Med J. 1996 Dec;72(854):731-8. doi: 10.1136/pgmj.72.854.731. PMID 9015466
- [Background] Cregler LL. Antithrombotic therapy in left ventricular thrombosis and systemic embolism. Am Heart J. 1992 Apr;123(4 Pt 2):1110-4. doi: 10.1016/0002-8703(92)91069-d. PMID 1553880